CLINICAL TRIAL: NCT00611767
Title: Gamma-Aminobutyric Acid (GABA) Mechanisms Underlying the Vulnerability to Alcohol Dependence
Brief Title: GABA Mechanisms Underlying the Vulnerability to Alcohol Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 0510000664; VA Merit Grant
Record Dates: First submitted 2007-12-27; First posted 2008-02-11 (Estimated); Results first posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2016-11

CONDITIONS: Alcoholism
Keywords: Thiopental; Alcohol; Family History; Vulnerability; GABA
MeSH Terms: conditions — Alcoholism | interventions — Thiopental

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family History Negative for Alcoholism (Active Comparator): Family History Negative for Alcoholism subjects will receive 2 interventions
  Interventions: Drug: Thiopental
- Family History Positive for Alcoholism (Placebo Comparator): Family History Positive for Alcoholism subjects will receive 2 interventions
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Thiopental — A 2-day test design involving 2 conditions: saline (Placebo) or Thiopental 1.5mg/kg (loading) with a subsequent infusion rate of 40 mcg/kg/minute (60 minute infusion).
  Arms: Family History Negative for Alcoholism
Drug: Placebo — A 2-day test design involving 2 conditions: saline (Placebo) or Thiopental 1.5mg/kg (loading) with a subsequent infusion rate of 40 mcg/kg/minute (60 minute infusion).
  Arms: Family History Positive for Alcoholism

SUMMARY:
This Project will explore the hypothesis that individuals with a family history positive for alcohol dependence (without any current Axis I disorder, except nicotine dependence), experience an alteration in the reward "valence" (balance of positive and negative effects) of the GABAA receptor agonist barbiturate (thiopental) compared to family history negative age-matched subjects. Further, variation in genes involved in brain GABA function may influence the risk for alcoholism by altering a component of the discriminative stimulus effects of ethanol.

DETAILED DESCRIPTION:
This project will explore the hypothesis that individuals with a family history positive for alcohol dependence (FHP) (without any current DSM-IV Axis I disorder, except nicotine dependence), experience an alteration in the reward "valence" (balance of positive and negative effects) of the GABA-A receptor agonist barbiturate (thiopental) compared to family history negative (FHN) age-matched subjects. Further, the effect of variations in genes important in regulating brain GABA function may alter a component of the discriminative stimulus effects of ethanol. FHP individuals are defined as individuals with at least one first-degree relative and another first- or second-degree relatives. Preliminary results suggest that FHP individuals showed an attenuated response to thiopental as measured by the descending limb of the BAES during thiopental infusion relative to the FHN group. Further, preliminary results suggest that variation in genes involved in brain GABA function, glutamate decarboxylase-65 (GAD65), may influence the risk for alcoholism by altering a component of the discriminative stimulus effects of ethanol.

We plan to recruit 2 groups of healthy subjects between the ages of 21-30, one with a family history of alcoholism (family history positive=FHP) and a sex-matched control group without a family history of alcoholism (family history negative=FHN), to undergo two test days scheduled 3 days apart, in a randomized double-blind fashion. Test days will involve a 60-minute intravenous infusion of each of 2 conditions: saline or thiopental, in a randomized order under double-blind conditions. Behavioral ratings include the Biphasic Alcohol Effects Scale (BAES) and Visual Analog Scales (VAS). Exploratory measures include event-related potential recordings (ERP) and measures of eye-to-hand coordination. Blood will be collected for Deoxyribonucleic acid (DNA) extraction and genotyping.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female between the ages of 21 and 30 years
2. medically and neurologically healthy on the basis of history, physical examination, Electrocardiogram (EKG), screening laboratories
3. absence of any evidence of substance abuse (with the exception of nicotine dependence) on the basis of history and drug and ethanol-free at the time of testing based on urine toxicology and breath alcohol levels at screening and on each test day.

Exclusion Criteria:

1. Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) Axis I psychiatric and substance abuse or dependence diagnosis by history on psychiatric evaluation that includes a structured diagnostic interview (SCID)
2. unwillingness to remain alcohol-free for three days prior to each test day;
3. for women, positive pregnancy test at screening or intention to engage in unprotected sex during the study and
4. alcohol naive. For Family History Positive Subjects: 1) Biological father and another first or second-degree biological relative with history of alcoholism by Family History Assessment Module (FHAM) developed by The Collaborative Study on the Genetics of Alcoholism (COGA).

For Family History Negative Subjects: NO family history of alcoholism in any first or second-degree relatives. Subjects must reliably report on three first-degree relatives.

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2005-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ismene L Petrakis, MD, Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

REFERENCES:
- [Result] Petrakis IL, Kerfoot K, Pittman B, Perrino A, Koretski J, Newcomb J, Limoncelli D, Acampora G, Ralevski E. Subjective Effects of Thiopental in Young Adults with and without a Family History of Alcoholism. J Addict Res Ther. 2012 May 14;Suppl 7(2):6336. doi: 10.4172/2155-6105.S7-002. PMID 24273687

RESULTS

PARTICIPANT FLOW:
Groups:
- Family History Negative for Alcoholism: Male or female (post-menopausal, surgically sterile, or negative pregnancy test at screening and agreement to utilize an established birth control during the testing period) between the age of 21 and 30 yrs, medically healthy, who have been absence of any evidence of substance abuse (with the exception of nicotine dependence) diagnosis by the non-patient version of the structured clinical interview (SCID). No family history of alcoholism in any first or second-degree relatives.
- Family History Positive for Alcoholism: Male or female (post-menopausal, surgically sterile, or negative pregnancy test at screening and agreement to utilize an established birth control during the testing period) between the age of 21 and 30 yrs, medically healthy, who have been absence of any evidence of substance abuse (with the exception of nicotine dependence) diagnosis by the non-patient version of the structured clinical interview (SCID). Biological father and another first or second-degree biological relative with a history of alcoholism by Family History Assessment Module (FHAM) developed by The Collaborative Study on the Genetics of Alcoholism (COGA).
Period: Overall Study
Arm/Group | Family History Negative for Alcoholism | Family History Positive for Alcoholism
Started | 49 | 24
Thiopental Test Day | 3 | 1
Placebo Test Day | 6 | 1
Completed | 40 | 22
Not Completed | 9 | 2
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Thiopental not available | 3 | 0
Not completed — didn't like the medication | 1 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Family History Positive for Alcoholism: Male or female (post-menopausal, surgically sterile, or negative pregnancy test at screening and agreement to utilize an established birth control during the testing period) between the age of 21 and 30 yrs, medically healthy, who have been absence of any evidence of substance abuse (with the exception of nicotine dependence) diagnosis by the non-patient version of the structured clinical interview (SCID). Biological father and another first or second-degree biological relative with a history of alcoholism by Family History Assessment Module (FHAM) developed by COGA.
- Total: Total of all reporting groups
Arm/Group | Family History Negative for Alcoholism | Family History Positive for Alcoholism | Total
Number analyzed (Participants) | 49 | 24 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 24 | 73
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.02 (2.5) | 24.63 (3.06) | 24.22 (2.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 10 | 35
  Male | 24 | 14 | 38
Region of Enrollment [Number; unit: participants]
  United States | 49 | 24 | 73

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scales of Similarity to Alcohol - Baseline
Description: Visual Analog Scale of Similarity to Alcohol data using the Likert scale (0 Not at all similar to alcohol - 7 Extremely similar to alcohol) evaluating the similarity of drug effects to alcohol
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Family History Positive: Family History Positive for Alcoholism subjects will receive 2 interventions
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 0 (0) | 0 (0)
  Placebo | 0 (0) | 0 (0)

2. Primary Outcome: Visual Analog Scales of Similarity to Alcohol - 15 Minutes
Description: as for outcome 1
Time Frame: 15 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 3.23 (2.08) | 2.35 (1.90)
  Placebo | 0.04 (0.30) | 0.17 (0.65)

3. Primary Outcome: Visual Analog Scales of Similarity to Alcohol - 45 Minutes
Description: as for outcome 1
Time Frame: 45 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 2.91 (1.97) | 1.87 (1.71)
  Placebo | 0.04 (0.21) | 0.04 (0.21)

4. Primary Outcome: Visual Analog Scales of Similarity to Alcohol - 80 Minutes
Description: as for outcome 1
Time Frame: 80 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 22
  Thiopental | 0.84 (1.33) | 0.50 (0.74)
  Placebo | 0.04 (0.30) | 0 (0)

5. Primary Outcome: Visual Analog Scales of Similarity to Alcohol - 110 Minutes
Description: as for outcome 1
Time Frame: 110 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 0.35 (0.92) | 0.22 (0.85)
  Placebo | 0.11 (0.74) | 0 (0)

6. Primary Outcome: Visual Analog Scales of Similarity to Alcohol - 170 Minutes
Description: as for outcome 1
Time Frame: 170 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 0.02 (0.15) | 0 (0)
  Placebo | 0.02 (0.15) | 0 (0)

7. Primary Outcome: Visual Analog Scales of Similarity to Alcohol - 230 Minutes
Description: as for outcome 1
Time Frame: 230 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 0 (0) | 0 (0)
  Placebo | 0 (0) | 0 (0)

8. Secondary Outcome: Number of Drinks Felt Consumed at Baseline
Description: The Number of Drinks Scale asks Subjects to report on the number of alcoholic drinks they felt they had consumed.
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: number of drinks felt consumed
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
number of drinks felt consumed
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 0 (0) | 0 (0)
  Placebo | 0 (0) | 0 (0)

9. Secondary Outcome: Number of Drinks Felt Consumed - 15 Minutes
Description: The Number of Drinks Scale asks Subjects to report on the number of alcoholic drinks they felt they had consumed.
Time Frame: 15 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: number of drinks felt consumed
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
number of drinks felt consumed
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 3.28 (2.10) | 3.22 (2.63)
  Placebo | 0.11 (0.43) | 0.17 (0.49)

10. Secondary Outcome: Number of Drinks Felt Consumed - 45 Minutes
Description: The Number of Drinks Scale asks Subjects to report on the number of alcoholic drinks they felt they had consumed.
Time Frame: 45 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: number of drinks felt consumed
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
number of drinks felt consumed
  Thiopental: number analyzed (Participants) | 38 | 22
  Thiopental | 3 (2) | 2.91 (2.67)
  Placebo: number analyzed (Participants) | 40 | 23
  Placebo | 0.03 (0.16) | 0.04 (0.21)

11. Secondary Outcome: Number of Drinks Felt Consumed - 80 Minutes
Description: The Number of Drinks Scale asks Subjects to report on the number of alcoholic drinks they felt they had consumed.
Time Frame: 80 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: number of drinks felt consumed
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
number of drinks felt consumed
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 1.14 (1.78) | 0.96 (1.15)
  Placebo | 0.04 (0.30) | 0 (0)

12. Secondary Outcome: Number of Drinks Felt Consumed - 110 Minutes
Description: The Number of Drinks Scale asks Subjects to report on the number of alcoholic drinks they felt they had consumed.
Time Frame: 110 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: number of drinks felt consumed
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
number of drinks felt consumed
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 0.35 (0.92) | 0.22 (0.6)
  Placebo | 0.04 (0.30) | 0 (0)

13. Secondary Outcome: Number of Drinks Felt Consumed - 170 Minutes
Description: The Number of Drinks Scale asks Subjects to report on the number of alcoholic drinks they felt they had consumed.
Time Frame: 170 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: number of drinks felt consumed
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
number of drinks felt consumed
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 0 (0) | 0 (0)
  Placebo | 0.02 (0.15) | 0 (0)

14. Secondary Outcome: Number of Drinks Felt Consumed - 230 Minutes
Description: The Number of Drinks Scale asks Subjects to report on the number of alcoholic drinks they felt they had consumed.
Time Frame: 230 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: number of drinks felt consumed
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
number of drinks felt consumed
  Thiopental: number analyzed (Participants) | 41 | 23
  Thiopental | 0 (0) | 0 (0)
  Placebo | 0 (0) | 0 (0)

15. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Stimulant - Baseline
Description: Self-report rating scale used to measure stimulant effects (0 not at all stimulated - 70 extremely stimulated)
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 1.86 (4.41) | 1.22 (3.67)
  Placebo | 2.74 (7.16) | 1.91 (5.73)

16. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Stimulant - 15 Minutes
Description: Self-report rating scale used to measure stimulant effects (0 not at all stimulated - 70 extremely stimulated)
Time Frame: 15 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 5.26 (9.38) | 3.87 (6.24)
  Placebo | 1.5 (3.97) | 1.87 (4.46)

17. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Stimulant - 45 Minutes
Description: Self-report rating scale used to measure stimulant effects (0 not at all stimulated - 70 extremely stimulated)
Time Frame: 45 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 2.33 (4.07) | 2.70 (4.99)
  Placebo | 1.13 (3.21) | 1.57 (3.72)

18. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Stimulant - 80 Minutes
Description: Self-report rating scale used to measure stimulant effects (0 not at all stimulated - 70 extremely stimulated)
Time Frame: 80 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 1.37 (2.82) | 1.78 (4.38)
  Placebo | 1.5 (4.21) | 1.35 (3.33)

19. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Stimulant- 110 Minutes
Description: Self-report rating scale used to measure stimulant effects (0 not at all stimulated - 70 extremely stimulated)
Time Frame: 110 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 1.12 (2.22) | 1.52 (3.94)
  Placebo | 1.44 (4.38) | 1.91 (4.80)

20. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Stimulant - 170 Minutes
Description: Self-report rating scale used to measure stimulant effects (0 not at all stimulated - 70 extremely stimulated)
Time Frame: 170 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 0.98 (2.33) | 1.39 (3.73)
  Placebo | 1.85 (6.16) | 1.65 (4.00)

21. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Stimulant - 230 Minutes
Description: Self-report rating scale used to measure stimulant effects (0 not at all stimulated - 70 extremely stimulated)
Time Frame: 230 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 1 (2.01) | 2.30 (6.32)
  Placebo | 1.72 (4.70) | 2.04 (5.17)

22. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Sedative Baseline
Description: Self-report rating scale used to measure sedative effects (0 not at all sedated - 70 extremely sedated)
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 1.49 (2.55) | 0.48 (0.95)
  Placebo | 1.20 (2.52) | 0.44 (1.31)

23. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Sedative - 15 Minutes
Description: Self-report rating scale used to measure sedative effects (0 not at all sedated - 70 extremely sedated)
Time Frame: 15 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 16.07 (17.75) | 6.74 (8.30)
  Placebo | 1.41 (3.29) | 2.04 (6.87)

24. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Sedative - 45 Minutes
Description: Self-report rating scale used to measure sedative effects (0 not at all sedated - 70 extremely sedated)
Time Frame: 45 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 15.83 (13.79) | 9.30 (12.10)
  Placebo | 1.70 (4.61) | 1.17 (3.94)

25. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Sedative - 80 Minutes
Description: Self-report rating scale used to measure sedative effects (0 not at all sedated - 70 extremely sedated)
Time Frame: 80 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 7.98 (10.34) | 3.48 (6.07)
  Placebo | 0.94 (2.27) | 0.74 (2.34)

26. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Sedative - 110 Minutes
Description: Self-report rating scale used to measure sedative effects (0 not at all sedated - 70 extremely sedated)
Time Frame: 110 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 2.37 (4.34) | 1.61 (4.33)
  Placebo | 0.63 (1.88) | 0.78 (2.59)

27. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Sedative - 170 Minutes
Description: Self-report rating scale used to measure sedative effects (0 not at all sedated - 70 extremely sedated)
Time Frame: 170 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 0.83 (1.87) | 0.52 (1.90)
  Placebo | 0.26 (0.74) | 0.44 (1.16)

28. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Sedative - 230 Minutes
Description: Self-report rating scale used to measure sedative effects (0 not at all sedated - 70 extremely sedated)
Time Frame: 230 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 0.45 (1.33) | 0.22 (0.85)
  Placebo | 0.15 (0.52) | 0.26 (0.75)

29. Secondary Outcome: Visual Analog Scales (VAS) - High - Baseline
Description: visual analog scale (VAS): self-report scale used to measure high (0 not at all High - 7 extremely High)
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 0 (0) | 0 (0)
  Placebo | 0 (0) | 0 (0)

30. Secondary Outcome: Visual Analog Scales (VAS) - High - 15 Minutes
Description: visual analog scale (VAS): self-report scale used to measure high (0 not at all High - 7 extremely High)
Time Frame: 15 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 2.35 (2.25) | 1.74 (1.66)
  Placebo | 0 (0) | 0 (0)

31. Secondary Outcome: Visual Analog Scales (VAS) - High - 45 Minutes
Description: visual analog scale (VAS): self-report scale used to measure high (0 not at all High - 7 extremely High)
Time Frame: 45 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 1.69 (1.80) | 1.26 (2.03)
  Placebo | 0 (0) | 0 (0)

32. Secondary Outcome: Visual Analog Scales (VAS) - High - 80 Minutes
Description: visual analog scale (VAS): self-report scale used to measure high (0 not at all High - 7 extremely High)
Time Frame: 80 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 0.40 (1.00) | 0.61 (1.08)
  Placebo | 0.02 (0.15) | 0 (0)

33. Secondary Outcome: Visual Analog Scales (VAS) - High - 110 Minutes
Description: visual analog scale (VAS): self-report scale used to measure high (0 not at all High - 7 extremely High)
Time Frame: 110 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 0.14 (0.64) | 0.13 (0.46)
  Placebo | 0 (0) | 0 (0)

34. Secondary Outcome: Visual Analog Scales (VAS) - High - 170 Minutes
Description: visual analog scale (VAS): self-report scale used to measure high (0 not at all High - 7 extremely High)
Time Frame: 170 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 0 (0) | 0 (0)
  Placebo | 0 (0) | 0 (0)

35. Secondary Outcome: Visual Analog Scales (VAS) - High - 230 Minutes
Description: visual analog scale (VAS): self-report scale used to measure high (0 not at all High - 7 extremely High)
Time Frame: 230 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 0 (0) | 0 (0)
  Placebo | 0 (0) | 0 (0)

36. Secondary Outcome: Visual Analog Scales (VAS) - Buzzed - Baseline
Description: visual analog scale (VAS): self-report scale used to measure buzzed (0 not at all buzzed - 7 extremely buzzed)
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 0 (0) | 0 (0)
  Placebo | 0 (0) | 0 (0)

37. Secondary Outcome: Visual Analog Scales (VAS) - Buzzed - 15 Minutes
Description: visual analog scale (VAS): self-report scale used to measure buzzed (0 not at all buzzed - 7 extremely buzzed)
Time Frame: 15 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 2.07 (2.06) | 1.65 (1.85)
  Placebo | 0 (0) | 0.04 (0.21)

38. Secondary Outcome: Visual Analog Scales (VAS) - Buzzed - 45 Minutes
Description: visual analog scale (VAS): self-report scale used to measure buzzed (0 not at all buzzed - 7 extremely buzzed)
Time Frame: 45 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 1.74 (1.78) | 1.26 (1.94)
  Placebo | 0 (0) | 0.04 (0.21)

39. Secondary Outcome: Visual Analog Scales (VAS) - Buzzed - 80 Minutes
Description: visual analog scale (VAS): self-report scale used to measure buzzed (0 not at all buzzed - 7 extremely buzzed)
  .
Time Frame: 80 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 0.21 (0.68) | 0.52 (0.99)
  Placebo | 0.04 (0.30) | 0 (0)

40. Secondary Outcome: Visual Analog Scales (VAS) - Buzzed - 110 Minutes
Description: visual analog scale (VAS): self-report scale used to measure buzzed (0 not at all buzzed - 7 extremely buzzed)
Time Frame: 110 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 0.02 (0.15) | 0.13 (0.46)
  Placebo | 0.02 (0.15) | 0 (0)

41. Secondary Outcome: Visual Analog Scales (VAS) - Buzzed - 170 Minutes
Description: visual analog scale (VAS): self-report scale used to measure buzzed (0 not at all buzzed - 7 extremely buzzed)
Time Frame: 170 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 0.02 (0.15) | 0 (0)
  Placebo | 0 (0) | 0 (0)

42. Secondary Outcome: Visual Analog Scales (VAS) - Buzzed - 230 Minutes
Description: visual analog scale (VAS): self-report scale used to measure buzzed (0 not at all buzzed - 7 extremely buzzed)
Time Frame: 230 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 0 (0) | 0 (0)
  Placebo | 0 (0) | 0 (0)

43. Secondary Outcome: Visual Analog Scales (VAS) - Drowsy - Baseline
Description: visual analog scale (VAS): self-report scale used to measure drowsy (0 not at all drowsy - 7 extremely drowsy)
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 0.61 (1.05) | 0.52 (1.04)
  Placebo | 0.22 (0.51) | 0.48 (1.31)

44. Secondary Outcome: Visual Analog Scales (VAS) - Drowsy - 15 Minutes
Description: visual analog scale (VAS): self-report scale used to measure drowsy (0 not at all drowsy - 7 extremely drowsy)
Time Frame: 15 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 2.86 (2.48) | 1.74 (1.86)
  Placebo | 0.39 (0.71) | 0.35 (0.57)

45. Secondary Outcome: Visual Analog Scales (VAS) - Drowsy - 45 Minutes
Description: visual analog scale (VAS): self-report scale used to measure drowsy (0 not at all drowsy - 7 extremely drowsy)
  .
Time Frame: 45 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 3.02 (2.44) | 2.74 (2.01)
  Placebo | 0.44 (0.91) | 0.39 (0.58)

46. Secondary Outcome: Visual Analog Scales (VAS) - Drowsy - 80 Minutes
Description: visual analog scale (VAS): self-report scale used to measure drowsy (0 not at all drowsy - 7 extremely drowsy)
Time Frame: 80 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 2.14 (1.82) | 1.48 (1.59)
  Placebo | 0.20 (0.45) | 0.35 (0.78)

47. Secondary Outcome: Visual Analog Scales (VAS) - Drowsy - 110 Minutes
Description: visual analog scale (VAS): self-report scale used to measure drowsy (0 not at all drowsy - 7 extremely drowsy)
Time Frame: 110 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 1.19 (1.64) | 1.13 (1.25)
  Placebo | 0.13 (0.4) | 0.30 (0.70)

48. Secondary Outcome: Visual Analog Scales (VAS) - Drowsy - 170 Minutes
Description: visual analog scale (VAS): self-report scale used to measure drowsy (0 not at all drowsy - 7 extremely drowsy)
Time Frame: 170 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 0.38 (0.66) | 0.26 (0.54)
  Placebo | 0.15 (0.56) | 0.22 (0.60)

49. Secondary Outcome: Visual Analog Scales (VAS) - Drowsy - 230 Minutes
Description: visual analog scale (VAS): self-report scale used to measure drowsy (0 not at all drowsy - 7 extremely drowsy)
Time Frame: 230 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 0.31 (0.60) | 0.13 (0.34)
  Placebo | 0.11 (0.43) | 0.17 (0.58)

50. Secondary Outcome: Visual Analog Scales (VAS) - Depressed - Baseline
Description: visual analog scale (VAS): self-report scale used to measure depressed (0 not at all depressed - 7 extremely depressed)
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 0.07 (0.34) | 0.04 (0.21)
  Placebo | 0 (0) | 0 (0)

51. Secondary Outcome: Visual Analog Scales (VAS) - Depressed - 15 Minutes
Description: visual analog scale (VAS): self-report scale used to measure depressed (0 not at all depressed - 7 extremely depressed)
Time Frame: 15 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 0.02 (0.15) | 0.13 (0.63)
  Placebo | 0.04 (0.30) | 0 (0)

52. Secondary Outcome: Visual Analog Scales (VAS) - Depressed - 45 Minutes
Description: visual analog scale (VAS): self-report scale used to measure depressed (0 not at all depressed - 7 extremely depressed)
Time Frame: 45 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 0.02 (0.15) | 0.09 (0.42)
  Placebo | 0.04 (0.30) | 0 (0)

53. Secondary Outcome: Visual Analog Scales (VAS) - Depressed - 80 Minutes
Description: visual analog scale (VAS): self-report scale used to measure depressed (0 not at all depressed - 7 extremely depressed)
Time Frame: 80 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 0.02 (0.15) | 0.04 (0.21)
  Placebo | 0 (0) | 0 (0)

54. Secondary Outcome: Visual Analog Scales (VAS) - Depressed - 110 Minutes
Description: visual analog scale (VAS): self-report scale used to measure depressed (0 not at all depressed - 7 extremely depressed)
Time Frame: 110 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 0 (0) | 0 (0)
  Placebo | 0 (0) | 0 (0)

55. Secondary Outcome: Visual Analog Scales (VAS) - Depressed - 170 Minutes
Description: visual analog scale (VAS): self-report scale used to measure depressed (0 not at all depressed - 7 extremely depressed)
Time Frame: 170 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 0 (0) | 0 (0)
  Placebo | 0 (0) | 0 (0)

56. Secondary Outcome: Visual Analog Scales (VAS) - Depressed - 230 Minutes
Description: visual analog scale (VAS): self-report scale used to measure depressed (0 not at all depressed - 7 extremely depressed)
Time Frame: 230 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 0.02 (0.15) | 0 (0)
  Placebo | 0 (0) | 0 (0)

57. Secondary Outcome: Visual Analog Scales (VAS) - Anxious - Baseline
Description: visual analog scale (VAS): self-report scale used to measure anxiety (0 not at all anxious - 7 extremely anxious)
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 0.12 (0.45) | 0.13 (0.34)
  Placebo | 0.09 (0.29) | 0.13 (0.34)

58. Secondary Outcome: Visual Analog Scales (VAS) - Anxious - 15 Minutes
Description: visual analog scale (VAS): self-report scale used to measure anxiety (0 not at all anxious - 7 extremely anxious)
Time Frame: 15 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 0.21 (0.89) | 0.22 (0.85)
  Placebo | 0 (0) | 0.04 (0.21)

59. Secondary Outcome: Visual Analog Scales (VAS) - Anxious - 45 Minutes
Description: visual analog scale (VAS): self-report scale used to measure anxiety (0 not at all anxious - 7 extremely anxious)
Time Frame: 45 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 0.07 (0.34) | 0.13 (0.46)
  Placebo | 0 (0) | 0 (0)

60. Secondary Outcome: Visual Analog Scales (VAS) - Anxious - 80 Minutes
Description: visual analog scale (VAS): self-report scale used to measure anxiety (0 not at all anxious - 7 extremely anxious)
Time Frame: 80 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 0.05 (0.31) | 0 (0)
  Placebo | 0 (0) | 0.04 (0.21)

61. Secondary Outcome: Visual Analog Scales (VAS) - Anxious - 110 Minutes
Description: visual analog scale (VAS): self-report scale used to measure anxiety (0 not at all anxious - 7 extremely anxious)
Time Frame: 110 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 0 (0) | 0 (0)
  Placebo | 0.02 (0.15) | 0 (0)

62. Secondary Outcome: Visual Analog Scales (VAS) - Anxious - 170 Minutes
Description: visual analog scale (VAS): self-report scale used to measure anxiety (0 not at all anxious - 7 extremely anxious)
Time Frame: 170 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 0 (0) | 0 (0)
  Placebo | 0.04 (0.30) | 0.04 (0.21)

63. Secondary Outcome: Visual Analog Scales (VAS) - Anxious - 230 Minutes
Description: visual analog scale (VAS): self-report scale used to measure anxiety (0 not at all anxious - 7 extremely anxious)
Time Frame: 230 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 0 (0) | 0.04 (0.21)
  Placebo | 0 (0) | 0.04 (0.21)

64. Secondary Outcome: Clinician Administered Dissociative Symptoms Scale - Patient Rated - Baseline
Description: Clinician Administered Dissociative Symptoms Scale (CADSS) is a patient and Clinician rated measurement of dissociative states induced by thiopental (0 not at all dissociative - 84 extreme dissociative)
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 44 | 23
  Thiopental | 0 (0) | 0 (0)
  Placebo | 0 (0) | 0 (0)

65. Secondary Outcome: Clinician Administered Dissociative Symptoms Scale - Patient Rated - 15 Minutes
Description: as for outcome 64
Time Frame: 15 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 44 | 23
  Thiopental | 2.57 (3.35) | 1.74 (1.79)
  Placebo | 0.02 (0.15) | 0.04 (0.21)

66. Secondary Outcome: Clinician Administered Dissociative Symptoms Scale - Patient Rated - 80 Minutes
Description: as for outcome 64
Time Frame: 80 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 44 | 23
  Thiopental | 0.73 (1.58) | 0.83 (1.56)
  Placebo | 0 (0) | 0 (0)

67. Secondary Outcome: Clinician Administered Dissociative Symptoms Scale - Patient Rated - 110 Minutes
Description: as for outcome 64
Time Frame: 110 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 44 | 23
  Thiopental | 0.43 (1.59) | 0.22 (0.42)
  Placebo | 0 (0) | 0 (0)

68. Secondary Outcome: Clinician Administered Dissociative Symptoms Scale - Clinician Rated - Baseline
Description: Clinician Administered Dissociative Symptoms Scale (CADSS) is a patient and Clinician rated measurement of dissociative states induced by thiopental (0 not at all dissociative - 20 extreme dissociative)
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 44 | 23
  Thiopental | 0.02 (0.15) | 0 (0)
  Placebo | 0 (0) | 0 (0)

69. Secondary Outcome: Clinician Administered Dissociative Symptoms Scale - Clinician Rated - 15 Minutes
Description: as for outcome 68
Time Frame: 15 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 44 | 23
  Thiopental | 1.43 (2.39) | 1.04 (1.72)
  Placebo | 0.02 (0.15) | 0 (0)

70. Secondary Outcome: Clinician Administered Dissociative Symptoms Scale - Clinician Rated - 80 Minutes
Description: as for outcome 68
Time Frame: 80 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 44 | 23
  Thiopental | 0.68 (1.54) | 0.35 (0.65)
  Placebo | 0 (0) | 0.09 (0.42)

71. Secondary Outcome: Clinician Administered Dissociative Symptoms Scale - Clinician Rated - 110 Minutes
Description: as for outcome 68
Time Frame: 110 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
units on a scale
  Thiopental: number analyzed (Participants) | 44 | 23
  Thiopental | 0.21 (0.67) | 0.17 (0.49)
  Placebo | 0 (0) | 0 (0)

72. Secondary Outcome: Pegboard Task - Baseline (Dominant Hand)
Description: The pegboard task is a measure of coordination that measures reaction time; how long a subject takes to insert pegs into a pegboard puzzle, first using their dominant hand then using their non-dominant hand. A quicker time indicates greater coordination. Scores are timed in seconds
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
seconds
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 58.49 (9.39) | 60.57 (10.56)
  Placebo | 57.37 (6.84) | 60.78 (7.59)

73. Secondary Outcome: Pegboard Task - 15 Minutes (Dominant Hand)
Description: as for outcome 72
Time Frame: 15 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
seconds
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 84.56 (22.92) | 82.04 (16.36)
  Placebo | 65.11 (10.04) | 69.61 (13.68)

74. Secondary Outcome: Pegboard Task - Baseline (Non-Dominant Hand)
Description: as for outcome 72
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
seconds
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 64.19 (10.15) | 66.52 (10.95)
  Placebo | 62.98 (8.29) | 69.83 (13.21)

75. Secondary Outcome: Pegboard Task - 15 Minutes (Non-Dominant Hand)
Description: as for outcome 72
Time Frame: 15 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
seconds
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 91.19 (23.23) | 87.09 (19.99)
  Placebo | 71.13 (12.57) | 75.48 (13.74)

76. Secondary Outcome: Hopkins Verbal Learning Task (HVLT) - Total Recall
Description: Hopkins Verbal Learning Task (HVLT) - measures verbal memory and hippocampus function based on word recall. (0 = no words recalled - 36 = all words recalled)
Time Frame: 15 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: words recalled
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
words recalled
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 25.88 (6.14) | 26.96 (4.41)
  Placebo | 29.02 (3.94) | 29.35 (3.80)

77. Secondary Outcome: Hopkins Verbal Learning Task (HVLT) - Delayed Recall
Description: Hopkins Verbal Learning Task (HVLT) - measures verbal memory and hippocampus function with word recall at 30 minutes) (0 no words recalled - 12 all words recalled)
Time Frame: 45 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: words recalled
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
words recalled
  Thiopental: number analyzed (Participants) | 42 | 23
  Thiopental | 8.29 (3.39) | 8.74 (3.24)
  Placebo | 10.44 (1.75) | 10.04 (2.08)

78. Secondary Outcome: Verbal Fluency
Description: Verbal Fluency Task: requires subjects to generate as many words as possible beginning with a single letter (e.g., "H") during a one-minute interval. (total words in one-minute interval)
Time Frame: 15 minutes
Population: All available data was utilized in the analysis using mixed models.
Measure: Mean (Standard Deviation); unit: number of words
Arm/Group | Family History Negative for Alcoholism | Family History Positive
Number analyzed (Participants) | 46 | 23
number of words
  Thiopental: number analyzed (Participants) | 43 | 23
  Thiopental | 13.47 (4.11) | 13.96 (3.34)
  Placebo | 14.35 (4.42) | 14.04 (3.23)

ADVERSE EVENTS:
Description: There were no adverse events in this trial, so events are not listed separately for each intervention but are reported by trial arm.
Arm/Group | Family History Negative for Alcoholism | Family History Positive for Alcoholism
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/24
Other Adverse Events (participants affected / at risk) | 0/49 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes